CLINICAL TRIAL: NCT02384967
Title: Phase II Trial Assessing the Efficacy of a Reduced Dose Strategy of Darunavir to 400 mg/d in HIV-1 Infected Patients Virologically Suppressed Under a Once Daily Regimen Including Darunavir 800 mg/d and Two Nucleoside Reverse Transcriptase Inhibitors (NRTI), to Maintain the Viral Load Lower Than 50 Copies / mL at 48 Weeks of Treatment
Brief Title: Evaluation of a Dose Reduction of Darunavir (400 mg/d) in Virologically Suppressed HIV-1 Patients
Acronym: DARULIGHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 165 DARULIGHT
Record Dates: First submitted 2015-02-23; First posted 2015-03-10 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: HIV INFECTION
MeSH Terms: conditions — HIV Infections | interventions — Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Darunavir 400mg/d (Experimental): Tri-therapy containing Darunavir at dose of 400 mg/d.
  Interventions: Drug: Darunavir

INTERVENTIONS:
Drug: Darunavir — to assess efficacy of a reduced dose strategy of darunavir to 400 mg/d in HIV-1 infected patients virologically suppressed under a once daily regimen including darunavir 800 mg/d and two nucleoside reverse transcriptase inhibitors (NRTI), to maintain the viral load lower than 50 copies / mL at 48 weeks of treatment.
  Other Names: Prezista

SUMMARY:
Phase II trial assessing the efficacy of a reduced dose strategy of darunavir to 400 mg/d in HIV-1 infected patients virologically suppressed under a once daily regimen including darunavir 800 mg/d and two nucleoside reverse transcriptase inhibitors (NRTI), to maintain the viral load lower than 50 copies / mL at 48 weeks of treatment.

DETAILED DESCRIPTION:
Principal objective: To evaluate the proportion of subjects virologically suppressed at week 48 (viral load=VL ≤ 50 cp/mL) under a tri-therapy containing the darunavir at the dose of 400 mg/d.

Secondary objectives: To evaluate between baseline and week 48: proportions of subjects: in virological failure (confirmed VL > 50 cp/mL) confirmed by a 2nd measure made between 2 to 4 weeks, with VL ≤ 50 cp/mL and between 20 and 50 cp/mL, emerging drug resistance if virological failure, CD4 cell count evolution, HIV DNA evolution, morphological and glucido-lipid parameters modifications, digestive treatment tolerance , adherence to treatment, overall cost of antiretroviral therapy, factors associated to virological failure including baseline and nadir CD4 cell count, darunavir plasma level, baseline HIV DNA viral load.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults,
* age ≥ 18 years,
* with a once-a-day ritonavir-boosted darunavir 800mg/j containing regimen plus 2 NRTI (≥ 6 months),
* virologically controlled (VL ≤ 50 cp/ml,
* ≥ 1 year,
* at least 2 VL spaced at least 3 months apart in the last 12 months) CD4 count ≥ 300/mm3 ≥ 6 months,
* virus sensible to darunavir and the used NRTI (pretreatment resistance genotypic test available) and
* with no history of virological failure (VL > 200 cp/mL after ≥ 6 months under PI and/or used NRTI),
* no current opportunistic infection,
* renal clearance ≥ 60 mL/min if tenofovir is used,
* transaminases (SGOT, SGPT) plasma levels < 2N,
* hemoglobin > 11 g/dL,
* platelets count > 150 000/mm3,
* negative pregnancy test in women with childbearing potential,
* informed written consent signed by both the investigator and the subject,
* national insurance scheme (article L1121-11 of the French Public Health code),
* no participation to any other clinical trial

Exclusion Criteria:

* HIV-2 infection,
* current antiretroviral therapy different from a once-a-day ritonavir-boosted darunavir 800mg/j containing regimen plus 2 NRTI,
* virus genotypically resistant to darunavir and the used NRTIs,
* history of virological failure (VL > 200 cp/mL after ≥ 6 months under PI and/or used NRTI),
* irregular follow-up and/or history of lack of adherence to ART ≤ 12 months,
* current pregnancy,
* current opportunistic infection,
* associated treatment containing one or more drugs interacting with hepatic cytochromes,
* any addictive behaviors (alcohol consumption, drugs …) likely to jeopardize the safety of the treatment and / or patient compliance and adherence to the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with therapeutic success, defined as no virological failure | Week 48
  Virological failure is defined as confirmed VL > 50 cp/mL and no change of the strategy

SECONDARY OUTCOMES:
Proportions of patients with virological failure (confirmed VL > 50 cp/ml) | Week 48
Proportions of patients with VL < 50 cp/ml | Week 12, Week 24, Week 36, Week 48
Proportions of patients with VL between 20 and 50 cp/ml | Week 12, Week 24, Week 36, Week 48
Change from baseline in blood CD4 cell count at week 12, week 24, week 36 and week 48 | Week 12, Week 24, Week 36, Week 48
Change from baseline in blood HIV DNA at week 48 | Week 48
Emerging drug resistance if virological failure | Week 48
Treatment adherence | Week 48
Change from baseline in blood lipids at week 24 and week 48 | Week 24 and Week 48
Change from baseline in glucose at week 24 and week 48 | Week 24 and Week 48
Treatment Digestive tolerance | Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Louis, Paris, France

REFERENCES:
- [Derived] Le MP, Chaix ML, Chevret S, Bertrand J, Raffi F, Gallien S, El Abbassi EMB, Katlama C, Delobel P, Yazdanpanah Y, Saillard J, Molina JM, Peytavin G; ANRS 165 DARULIGHT Study Group. Pharmacokinetic modelling of darunavir/ritonavir dose reduction (800/100 to 400/100 mg once daily) in a darunavir/ritonavir-containing regimen in virologically suppressed HIV-infected patients: ANRS 165 DARULIGHT sub-study. J Antimicrob Chemother. 2018 Aug 1;73(8):2120-2128. doi: 10.1093/jac/dky193. PMID 29905808